CLINICAL TRIAL: NCT01795079
Title: Boston-Harvard Burn Injury Model System: Cortical Modulation With Transcranial Direct Current Stimulation (tDCS) for Neuropathic Symptoms Following Burn Injury
Brief Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Neuropathic Symptoms Following Burn Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Felipe Fregni, Associate Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-p-001996
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Results first posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Burn Injury; Chronic Pain; Pruritus; Itching
Keywords: transcranial stimulation; direct current
MeSH Terms: conditions — Burns; Chronic Pain; Pruritus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tDCS (Experimental): Subjects will undergo 20 minutes active tDCS.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): Subjects will undergo 20 minutes of sham stimulation.
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Subjects will undergo 15 sessions of tDCS stimulation (either active or sham), 1x per day at 20 minutes per session.
  Other Names: 1x1 low-intensity direct current stimulator; Soterix Medical

SUMMARY:
The purpose of this study is to see the effects of transcranial direct current stimulation (tDCS) on the pain and itching associated with burn injury. This study is part of the Boston-Harvard Burn Model System. The investigators hypothesize that there will be a decrease in pain levels with active stimulation, when compared to sham stimulation, using a 3 week stimulation schedule- 2 weeks of stimulation (10 consecutive days) followed by 1 week of stimulation (5 consecutive days) after three follow up visits at 2, 4 and 8 weeks after initial course of stimulation. The subject will also have follow ups at 2, 4 and 8 weeks after the second course of stimulation.

If a subject receives sham during the experiment, he/she may enroll in an open-label portion of the study and receive 10 days of active stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Providing informed consent to participate in the study
* Age 18 or older
* Burn injury with pain and/or itch that is moderate to severe
* Burn injury occurring at least 3 weeks prior to enrollment

Exclusion Criteria:

* Subjects with burns in scalp in the area of electrode placement
* Psychiatric disorders that have led to hospitalization within the past 6 months or signs of suicidality
* Learning disorders that may prevent patient's ability to complete assessments
* Unstable conditions preventing travel to study site
* Current use of any of the following anti-epileptic medications or dopaminergic medications known to reduce or inhibit the benefits of tDCS treatment: carbamazepine, oxcarbazepine, phenytoin
* Contraindications to tDCS including implanted metal plates in the head or implanted brain medical devices
* Pregnancy at time of enrollment
* History of other neurological conditions associated with structural anatomical changes (i.e. stroke, brain injury, Parkinson's)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-01; Primary Completion 2019-07 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD PhD MPH, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Boston-Harvard Burn Injury Model System Website — http://www.bh-bims.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Please note that 34 subjects consented to participated but 3 were screened out (after consent, there are additional tests to determine eligibility) and/or they dropped out before randomization (therefore, only 31 subjects were randomized).
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 16 | 15
Completed | 13 | 12
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (14) | 48 (14) | 48.5 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Scale
Description: Determine whether anodal transcranial direct current stimulation is effective in reducing pain in subjects with neuropathic pain due to burn injury, as measured by changes in the Brief Pain Inventory (BPI). Brief Pain Inventory (BPI) consist consists of a 9 part questionnaire. The questions include the severity of pain levels (worst, least, average, & current), the impact of pain on daily functioning in different areas (mood, walking, relationships, sleep, normal work, & general activity), current treatments and perceived effectiveness of current treatments. The VAS Pain scale is a simple 10- point scale (0 = ''no pain'', 10 = ''pain as bad as you can imagine'') measuring patients' worst pain and least pain, on average and at present time.
Time Frame: 2 weeks
Population: blinded assessment of scores at the primary endpoint (2 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 12
units on a scale | 4.45 (1.94) | 4.19 (1.45)

2. Primary Outcome: Change in Itch Severity/Activity Scale
Description: Determine whether anodal transcranial direct current stimulation is effective in reducing itch severity/activity in subjects with neuropathic itching due to burn injury, as measured by changes in the Visual Analog Scale (VAS) .This is a 0 to 10 scale, where 0 indicates no intensity and a 10 indicates unbearable intensity of itching.
Time Frame: 2 weeks
Population: blinded assessment at primary endpoint (2 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 12
units on a scale | 3.65 (2.91) | 1.83 (1.76)

3. Secondary Outcome: Change in Depression Scale
Description: Determine whether anodal transcranial direct current stimulation is effective in decreasing severity of depression in subjects with neuropathic pain and itching due to burn injury, as measured by changes in the Beck Depression Inventory (BDI). The Beck Depression Inventory (BDI) contains 21 questions, each answer being scored on a scale value of 0 to 3 (total from 0-63). Higher total scores indicate more severe depressive symptoms.
Time Frame: 2 weeks
Population: blinded assessment of scores at the primary endpoint (2 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 12
score on a scale | 9.1 (7.1) | 9.2 (7.8)

4. Secondary Outcome: Change in Post-Traumatic Stress Symptoms Scale
Description: Determine whether anodal transcranial direct current stimulation is effective in decreasing post-traumatic stress symptoms in subjects with neuropathic pain and itching due to burn injury, as measured by changes in the Impact of Event Scale Revised (IES-R).This 22-item scale is designed to measure severity of PTS symptoms associated with a traumatic event. Subjects rate their level of distress associated with the event on a 0-4 scale (0 means not at all distressed, 4 means extremely distressed). The IES-R yields a total score (ranging from 0 to 88) where higher scores represent higher stress
Time Frame: 2 weeks
Population: blinded assessment of scores at the primary endpoint(2 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 12
score on a scale | 10.8 (10.6) | 36.3 (16.5)

5. Secondary Outcome: Change in Anxiety Scale
Description: Determine whether anodal transcranial direct current stimulation is effective in decreasing severity of anxiety in subjects with neuropathic pain and itching due to burn injury, as measured by changes in the Visual Analog Scale (VAS).This is a self-evaluation scale that ranges from 0 to 10, where 0 means no anxiety and 10 means the worst anxiety ever.
Time Frame: 2 weeks
Population: blinded assessment at the primary endpoint (2 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 13 | 12
units on a scale | 3.25 (3.62) | 2.92 (3.37)

6. Other Pre Specified Outcome: Change in Quality of Life Scale
Description: Determine whether anodal transcranial direct current stimulation is effective in increasing quality of life in subjects with neuropathic pain and itching due to burn injury, as measured by changes in the Veterans RAND 36 Item Health Survey (VR-36). There are eight domains total including: bodily pain, role limitations due to physical problems, physical functioning, general health perception, vitality, social functioning, and role limitations due to mental health issues. Scores for each domain are from 0-100 with a higher score defining a more favorable health outcome.
Time Frame: 2 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Community Integration Scale
Description: Determine whether anodal transcranial direct current stimulation is effective in increasing community integration functional outcomes in subjects with neuropathic pain and itching due to burn injury, as measured by changes in the Community Integration Questionnaire (CIQ). Total CIQ scores were used as the outcome measure. Contains 15 itms assessing community integrations across three domains (Home integration, social integration, productive activity) . The total score can range from 0 to 29 points (0 - minimal integration to 29 -maximal integration). A positive change indicates an improvement in integration.
Time Frame: 2 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Period of stimulation (3 weeks)
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 2/16 | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS (N=16) | Sham tDCS (N=15)
Hedache (Nervous system disorders) | 2 (2) | 5 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT01795079/Prot_SAP_000.pdf